## INFORMED CONSENT FORM

## **Full Study Title:** Clinical and cost effectiveness of Alpha-Stim AID Cranial Electrotherapy Stimulations (CES); a naturalistic study in patients with a primary working diagnosis of moderate-to-severe generalised anxiety disorder who did not improve with low intensity psychological therapy intervention **Short Study Title:** Clinical and cost effectiveness of Alpha-Stim AID CES **Principal Investigator:** Dr Peter Caunt **Participant Study ID:** Please initial every box to indicate consent: 1. I confirm that I have read the information sheet dated 19 May 2016 version 1.0 for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. 2. I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. 3. I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from Electromedical Products International and The Microcurrent Site and authorised representatives, from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. 4. I understand that the information collected about me will be used to support other research in the future, and may be shared anonymously with other researchers.

6. I agree to take part in the above study.

5. I agree to my General Practitioner being informed of my participation in the study.

When completed: 1x copy for participant, 1x copy for investigator site file, 1x copy for the medical

record.